CLINICAL TRIAL: NCT06308601
Title: The Effect of Laughter Yoga on Loneliness, Anger and Salivary Cortisol Levels in Visually Impaired Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Arife Gur Boz, Nurse, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-12.1T/60
Record Dates: First submitted 2024-01-27; First posted 2024-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Nursing Caries; Laughter; Visual Impairment; Loneliness; Anger
Keywords: Visually impaired; Laughter Yoga; Nursing; Anger; Loneliness; Cortisol
MeSH Terms: conditions — Laughter; Vision Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Research Population: The population of this research is the visually impaired individuals who received service from the Disabled Department within the Ataturk Provincial Public Library in Konak district of Izmir province between 2023-2024.
  Research Sample: In the research, "G. Using the "Power-3.1.9.7" program, the sample size of the study was calculated at a 95% confidence level before the data collection phase. The standardized effect size was found to be 0.90 when calculated based on the mean and standard deviation values of previous studies. As a result, the minimum number of samples was calculated as 28 for each group with a 95% confidence level, 0.05 alpha value, 0.90 intervention effect size and 95% theoretical power. It is aimed to reach 56 people in total. Considering that there will be a 20% case loss in experimental studies in the literature (Pan, et al., 2019), the number of samples was determined as 60 (30 interventions; 30 controls).
Who Masked: Outcomes Assessor
Masking Description: Statistical evaluation of the research results will be made by an expert other than the researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): 8 sessions of laughter yoga will be applied to the experimental group.
  Interventions: Other: Laughter yoga
- control group (No Intervention): No application will be made to the control group. After the research is completed, laughter yoga can be applied by the researcher, at the request of the experimental group, within the framework of ethical responsibilities.

INTERVENTIONS:
Other: Laughter yoga — Laughter is an innate, most natural, sincere and universal response to humorous stimuli. Philosophically, it is explained by relief theory, conflict theory and superiority theory (Öztürk & Tezel, 2021). The emergence of laughter yoga was made by Dr., an Indian medical doctor, in 1995. It was created by combining breathing exercises and unconditional laughter with the work of Madan Kataria and his wife Madhuri Kataria. In laughter yoga, the individual can laugh in a simulated way with the interaction of group members, without a funny situation, joke or joke. The body cannot distinguish between real and unreal laughter, and fake laughter begins to turn into real laughter (Kataria, 2011).
  Arms: experimental group

SUMMARY:
Purpose: This project aimed to examine the effects of laughter yoga, which is accepted as an international nursing initiative, on loneliness, anger and salivary cortisol levels in visually impaired individuals. When the national and international literature was examined, no project was found that measured the results of laughter yoga as an intervention for visually impaired individuals. For this reason, planning an original project in this field aims to contribute to the literature. Thanks to the evidence obtained, laughter yoga, an innovative approach, can be disseminated in institutions and organizations serving visually impaired individuals as an evidence-based practice that can improve the social skills of individuals.

Scope and Target Audience: The project will be carried out with visually impaired individuals receiving services in the Disabled Persons Department within the Atatürk Provincial Public Library located in Konak district of Izmir. In this section, services are provided to 250 members who actively use the library and to visually impaired people from all over Turkey.

Method and Expected Result: The project was planned in a randomized controlled, pre-test post-test, single-blind follow-up consultancy design. With this initiative, a social rehabilitation environment will be provided for visually impaired individuals by taking an approach based on respect, understanding and awareness. Laughter yoga is expected to reduce the level of anger and loneliness in visually impaired individuals. At the same time, laughter yoga is expected to reduce cortisol levels, which are known to increase when faced with stress factors, and increase serotonin, which is associated with happiness and vitality, and endorphine, known as the body's natural painkiller. With laughter yoga sessions, a social environment will be created where visually impaired individuals will have an active and independent experience. Thanks to the expected evidence, laughter yoga can be popularized both in visually impaired individuals and in individuals with other disabilities. Within the scope of protecting and improving health, laughter yoga can be planned to be carried out as a routine nursing practice in disabled centers. Thus, by creating an environment where visually impaired individuals and nurses come together, a more accessible health service will be provided to individuals with special needs.

DETAILED DESCRIPTION:
The first scientist to study the effects of laughter on human health and physiological processes was Dr. William Fry. In his book "Anatomy of a Disease", Norman Cousins talks about the effect of laughter on pain. In the book; It is stated that "even morphine" does not help to sleep during the painful periods of ankylosing spondylitis disease, and 10 minutes of belly-waving laughter provides two hours of pain-free sleep. The emergence of laughter yoga was made by Dr., an Indian medical doctor, in 1995. It was created by combining breathing exercises and unconditional laughter with the work of Madan Kataria and his wife Madhuri Kataria. In laughter yoga, the individual can laugh in a simulated way with the interaction of group members, without a funny situation, joke or joke. The body cannot distinguish between real and unreal laughter, and fake laughter begins to turn into real laughter. Laughter yoga is used in many countries today. "Yoga" and "Laughter Yoga", which are frequently used in scientific studies, were added to the list of international nursing interventions by the authorities of the University of Iowa NIC (Nursing Interventions Classification) committee as two different interventions. The World Health Organization (WHO) reported the global strategy on the subject to the Seventy-Sixth World Health Assembly. In this report, traditional medicine is linked to Target 3 and Target 3.8 of the Sustainable Development Goals. These goals include promoting well-being and healthy living for everyone at all ages and access to quality primary health care while protecting against financial risks. The report draws attention to ways to integrate safe and evidence-based traditional and complementary medicine services into national and/or local health systems, especially at the primary care level, as appropriate, according to the national context and priorities. In the project, laughter yoga, a current approach to protecting and improving health, was chosen to be applied to visually impaired individuals as a low-risk, high-accessibility, potentially beneficial intervention for personal development.

Rapid population growth, aging and lifestyle changes will increase global demand for eye care in the coming years. WHO reported that as of 2019, at least 2.2 billion people worldwide have visual impairments. One billion of them have preventable visual impairment or a problem that has not yet been addressed. The report, prepared upon recommendation at the 70th World Health Assembly, examines inequalities in the scope and quality of prevention, treatment and rehabilitation services; It focuses on the lack of trained eye health service providers and the weak integration of eye care services into health systems, among others. In our country, there are conditions that restrict full and effective participation in society on equal terms with other individuals due to various levels of loss of physical, mental, spiritual and sensory abilities. An individual who is affected by attitudes and environmental conditions is defined as disabled. Disability by the Ministry of Family and Social Services of the Republic of Turkey; It is defined as a social phenomenon that affects all segments of society, regardless of economic and social status. Although approaches to people with disabilities vary across societies and cultures, today disability is no longer a problem that individuals and families have to deal with alone, but has become an issue that concerns the whole society. In this context, visually impaired individuals who are among disadvantaged groups and are at the center of global goals were determined as participants of the project.

In the project, one of the outcome measures in which laughter yoga was expected to have an effect on visually impaired individuals was determined as the level of loneliness. Lacking the power of sight means visually impaired; negative effects in physical, psychological and social aspects. Visually impaired people have the fear of living a life dependent on others, of not having a status in society, of encountering limitations in their interactions with other people, and of not being able to make friends. Compared to the general population, people with disabilities tend to have fewer friends, less social support, and are more socially isolated. Research conducted in England based on a nationally representative sample of approximately 17,000 working-age adults found that disabled people were significantly more likely to report loneliness than their non-disabled peers. According to the results of the same study, exposure to loneliness in visually impaired individuals is positively associated with the incidence and prevalence of mental health problems. In a study examining the relationship between disability and loneliness and including nine countries, disability was associated with a higher probability of loneliness. In a study conducted with visually impaired university students in China, it was stated that being visually impaired and self-stigma had a significant relationship with loneliness. There is increasing concern about the impact of restrictions imposed to control the COVID-19 pandemic, which has affected the world in recent years, on loneliness, especially in individuals with disabilities. In a study, it was stated that visually impaired individuals constantly experienced higher levels of loneliness during the pandemic. While loneliness remained relatively constant in individuals without disabilities, it increased in those with disabilities and especially those with visual impairments. In studies examining the effects of laughter yoga on loneliness, it has been stated that it reduces loneliness.

In the project, another outcome measure in which laughter yoga is expected to have an effect on visually impaired individuals was determined as the level of anger. The frustration, difficulties and perception of incomprehension that disabled individuals encounter while performing their daily life activities may cause their anger levels to increase. In a study conducted with visually impaired individuals, it was stated that the trait anger levels of the sample group were high, and men's trait anger score averages and anger expression mean scores were higher. In another study, anger levels were found to be higher in two separate groups, one with a visually impaired child and one with a mentally disabled child, compared to the group with a non-disabled child. According to the statements of caregivers of disabled individuals, the anger of 79.1% of disabled individuals increased during COVID-19. In order to strengthen the care provided to disabled individuals in our country, 'Behavior Shaping and Anger Management' training was given to approximately 150 personnel working in institutions providing boarding and day care services across the country. Emotion theorists have written that laughter relieves overly tense energy, improves social bonds, reduces distress, undoes negative emotions, and is closely associated with reducing anger. The expectation of visually impaired individuals from society is an approach based on respect, understanding and awareness, abandoning exclusionary, discriminatory and pity-oriented attitudes. Within the framework of this approach, while visually impaired individuals expect to be accepted as they are, they can increase their subjective well-being by participating in social, cultural and sports activities and socializing. WHO emphasizes that people with severe visual impairments have access to rehabilitation services that allow them to fully participate in society. It also recommends raising awareness and empowerment efforts that involve people and communities.

All important chemicals that help mood change, dopamine, oxytocin, serotonin and endorphins, which we call "happiness hormones", are released as a result of laughter. The strategic use of laughter in treatments is aimed at regulating emotions, creating emotional memories, establishing social bonds, reducing anxiety and alleviating social tension, and is associated with neural network bundles. In the study conducted with Korean university senior nursing students, 8 sessions of laughter therapy program, 60 minutes twice a week for 4 weeks, were applied to the participants who were under the stress of final exams and employment. There was a significant (p<0.001) improvement in salivary cortisol levels, subjective happiness and psychological stress of the students in the intervention group compared to the control group. There are studies showing that laughter yoga improves depressive symptoms, reduces levels of stress hormones and improves heart rate variability. In this context, cortisol, endorphin and serotonin values of visually impaired individuals will be taken into account to be used in measuring the project results, and this measurement will be carried out with a saliva test, which is an easy and harmless method.

ELIGIBILITY:
Inclusion Criteria:

* Receiving service from Izmir Ataturk Provincial Public Library
* Being visually impaired
* Volunteering to participate in the research.

Exclusion Criteria:

1. Those diagnosed with diabetes mellitus, hypertension, hypothyroidism, hyperaldosteronism, pregnancy, malignancy, congestive heart failure, psychotic disorder, chronic liver failure, nephrotic syndrome, chronic renal failure and those who are on continuous medication (Angiotensin converting enzyme inhibitors, angiotensin receptor blocker, phenytoin, barbiturate). Visually impaired individuals who use oral contraceptives, etc.) will be excluded from the scope as their salivary cortisol level may be affected.
2. Individuals with conditions for which laughter yoga is not recommended (having undergone abdominal surgery in the last three months, uncontrolled hypertension, glaucoma, hernia, epilepsy) will be excluded from the scope.

Exclusion criteria from the study: Not participating in any of the laughter yoga sessions, being newly diagnosed with diseases that may affect the cortisol level during the four-week period during which laughter yoga is performed, and conditions for which laughter yoga is not recommended are the exclusion criteria from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
salivary cortisol test | 1. test: 1 day before interventions 2.test: 1 day after interventions
  Saliva samples will be taken from the experimental group and control group and tested in the laboratory.
UCLA(University of California, Los Angeles) Loneliness Scale | 1. test: 1 day before interventions 2.test: 1 day after interventions
  The survey form will be read to visually impaired individuals and their answers will be marked and filled out.
  Rating: 4-point Likert (1 = I never experience it - 4 = I often experience it).
  Scale Scoring: Scores between 20-80 are taken from the scale. As the score increases, the level of loneliness increases.
Trait Anger Scale | 1. test: 1 day before interventions 2.test: 1 day after interventions
  The survey form will be read to visually impaired individuals and their answers will be marked and filled out.
  Rating: 4-point Likert (1 = never - 4 = always)
  Scale Scoring: The score that can be obtained from the scale varies between 10 and 40. As the score increases, the anger level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Gülengül Mermer, assoc. prof., Study Director — https://unisis.ege.edu.tr/researcher=gulengul.s.mermer
Locations (1):
- Ege University, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazdani M, Esmaeilzadeh M, Pahlavanzadeh S, Khaledi F. The effect of laughter Yoga on general health among nursing students. Iran J Nurs Midwifery Res. 2014 Jan;19(1):36-40. PMID 24554958
- [Background] Kuru Alici N, Zorba Bahceli P. Effects of Laughter Therapy on Life Satisfaction and Loneliness in Older Adults Living in Nursing Homes in Turkey: A Parallel Group Randomized Controlled Trial. Rehabil Nurs. 2021 Mar-Apr 01;46(2):104-112. doi: 10.1097/RNJ.0000000000000266. PMID 33646727
- [Background] Ozturk FO, Bayraktar EP, Tezel A. The effect of laughter yoga on loneliness, psychological resilience, and quality of life in older adults: A pilot randomized controlled trial. Geriatr Nurs. 2023 Mar-Apr;50:208-214. doi: 10.1016/j.gerinurse.2023.01.009. Epub 2023 Feb 15. PMID 36804028
- [Background] Kuru Alici N, Zorba Bahceli P, Emiroglu ON. The preliminary effects of laughter therapy on loneliness and death anxiety among older adults living in nursing homes: A nonrandomised pilot study. Int J Older People Nurs. 2018 Dec;13(4):e12206. doi: 10.1111/opn.12206. Epub 2018 Jul 13. PMID 30004172
- [Background] Lee JS, Lee SK. The Effects of Laughter Therapy for the Relief of Employment-Stress in Korean Student Nurses by Assessing Psychological Stress Salivary Cortisol and Subjective Happiness. Osong Public Health Res Perspect. 2020 Feb;11(1):44-52. doi: 10.24171/j.phrp.2020.11.1.07. PMID 32149041
- See also: Center for Nursing Classification and Clinical Effectiveness — http://nursing.uiowa.edu/cncce/nic-publications
- See also: WHO global report on traditional and complementary medicine 2019 — http://www.who.int/publications/i/item/978924151536
- See also: Global strategy on traditional medicine — http://apps.who.int/gb/ebwha/pdf_files/EB152/B152%2818%29-en.pdf
- See also: World report on vision — http://www.who.int/publications/i/item/world-report-on-vision